CLINICAL TRIAL: NCT01412333
Title: A Randomized, Double-Blind, Double-Dummy, Parallel-Group Study To Evaluate the Efficacy and Safety of Ocrelizumab in Comparison to Interferon Beta-1a (Rebif) in Patients With Relapsing Multiple Sclerosis
Brief Title: A Study of Ocrelizumab in Comparison With Interferon Beta-1a (Rebif) in Participants With Relapsing Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: WA21093; 2010-020315-36 (EudraCT Number)
Record Dates: First submitted 2011-08-08; First posted 2011-08-09 (Estimated); Results first posted 2017-07-18 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Relapsing Multiple Sclerosis
MeSH Terms: interventions — Interferon beta-1a; ocrelizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Interferon beta-1a 44 mcg SC (Active Comparator): Interferon beta-1a 44 mcg SC injections three times per week (with placebo infusions matching ocrelizumab infusions every 24 weeks).
  Interventions: Drug: Interferon beta-1a; Drug: Ocrelizumab-matching placebo
- Ocrelizumab (Experimental): Ocrelizumab 600 mg or matching placebo intravenous (IV) as 300 mg infusions on Days 1 and 15 for the first dose and as a single infusion of 600 mg for all subsequent infusions every 24 weeks, with placebo injections matching interferon beta-1a SC three times per week.
  Interventions: Drug: Ocrelizumab; Drug: Interferon beta-1a-matching placebo

INTERVENTIONS:
Drug: Interferon beta-1a
  Other Names: Rebif
  Arms: Interferon beta-1a 44 mcg SC
Drug: Ocrelizumab-matching placebo
  Arms: Interferon beta-1a 44 mcg SC
Drug: Ocrelizumab
  Other Names: RO4964913
  Arms: Ocrelizumab
Drug: Interferon beta-1a-matching placebo
  Arms: Ocrelizumab

SUMMARY:
This randomized, double-blind, double-dummy, parallel-group study will evaluate the efficacy and safety of ocrelizumab in comparison with interferon beta-1a (Rebif) in participants with relapsing multiple sclerosis. Participants will be randomized to receive either ocrelizumab 600 mg or matching placebo intravenous (IV) as 300 mg infusions on Days 1 and 15 for the first dose and as a single infusion of 600 mg for all subsequent infusions every 24 weeks, with placebo injections matching interferon beta-1a SC three times per week; or interferon beta-1a 44 mcg SC injections three times per week (with placebo infusions matching ocrelizumab infusions every 24 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of multiple sclerosis, in accordance with the revised McDonald criteria (2010)
* At least 2 documented clinical attacks within the last 2 years prior to screening or one clinical attack in the years prior to screening (but not within 30 days prior to screening)
* Neurologic stability for greater than or equal to (>/=) 30 days prior to both screening and baseline
* Expanded Disability Status Scale (EDSS) score 0 to 5.5 inclusive

Exclusion Criteria:

* Primary progressive multiple sclerosis
* Disease duration of more than 10 years in patients with EDSS score less than or equal to (</=) 2.0 at screening
* Contraindications for MRI
* Known presence of other neurological disorders which may mimic multiple sclerosis
* Pregnancy or lactation
* Requirement for chronic treatment with systemic corticosteroids or immunosuppressants during the course of the study
* History of or currently active primary or secondary immunodeficiency
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies
* Active infection, or history of or known presence of recurrent or chronic infection (for example, hepatitis B or C, Human Immunodeficiency Virus [HIV], syphilis, tuberculosis)
* History of progressive multifocal leukoencephalopathy
* Contraindications to or intolerance of oral or IV corticosteroids
* Contraindications to Rebif or incompatibility with Rebif use

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 835 (Actual)
Dates: Start 2011-09-20 (Actual); Primary Completion 2015-05-12 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (165):
- United States (48):
  - Hope Research Institute, Phoenix, Arizona
  - HonorHealth Neurology, Scottsdale, Arizona
  - Territory Neurology and Research Institute, Tucson, Arizona
  - Collaborative Neuroscience Research, LLC, Long Beach, California
  - Stanford University Medical Center, Palo Alto, California
  - University of Colorado, Denver, Colorado
  - Advanced Neurosciences Research LLC, Fort Collins, Colorado
  - Associated Neurologists of Southern CT PC, Fairfield, Connecticut
  - Infinity Clinical Research, Hollywood, Florida
  - University of Miami; Dept. of Neurology MS Center, Miami, Florida
  - Neurological Services of Orlando, Orlando, Florida
  - Lovelace Scientific Resources, Sarasota, Florida
  - University of South Florida, Tampa, Florida
  - Atlanta Neuroscience Institute, Atlanta, Georgia
  - Josephson Wallack Munshower Neurology PC, Indianapolis, Indiana
  - University of Kansas Medical Center, Kansas City, Kansas
  - MidAmerica Neuroscience Institute, Prairie Village, Kansas
  - Associates in Neurology PSC, Lexington, Kentucky
  - Dragonfly Research, LLC, Wellesley, Massachusetts
  - University of Massachusetts Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Wayne State University; Department of Neurology, Detroit, Michigan
  - The Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Holy Name Hospital, Teaneck, New Jersey
  - MS Comprehensive Care Center, Teaneck, New Jersey
  - Shore Neurology, Toms River, New Jersey
  - Empire Neurology, PC, Latham, New York
  - Weill Cornell MC-NY Presbyter; Dept. of Neurology/Neuroscience, Judith Jaffe Multiple Sclerosis Ctr, New York, New York
  - South Shore Neurologic Associates P.C., Patchogue, New York
  - University of Rochester Medical Center, Rochester, New York
  - SUNY at Stony Brook, Stony Brook, New York
  - The Neurological Institute PA, Charlotte, North Carolina
  - Neurology Associates PA, Hickory, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Columbus Neuroscience, Columbus, Ohio
  - Abington Neurological Associates, Abington, Pennsylvania
  - Absher Neurology PA, Greenville, South Carolina
  - Neurology Clinic PC, Cordova, Tennessee
  - Sibyl Wray MD Neurology PC, Knoxville, Tennessee
  - Advanced Neurosciences Institute, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Bhupesh Dihenia M.D. P.A., Lubbock, Texas
  - Central Texas Neurology Consultants, Round Rock, Texas
  - Integra Clinical Research, Llc, San Antonio, Texas
  - Neurology Center of San Antonio, San Antonio, Texas
  - Swedish Neuroscience Institute, Seattle, Washington
- Argentina (2):
  - ALPI-Inst. de Rehabilitacion Marcelo Fitte, Buenos Aires
  - STAT Research S.A., Ciudad de Buenos Airesa
- Belarus (4):
  - Grodno State Medical University, Hrodna, Grodnenskaya
  - Vitebsk; Regional Diagnostic Center, Vitebsk, Vitebsk Oblast
  - Vitebsk Regional Clinical Hospital, Vitebsk, Vitebsk Oblast
  - City Clinical Hospital #9, Minsk
- UZ Antwerpen, Edegem, Belgium
- Bosnia and Herzegovina (2):
  - University Clinic Ctr Sarajevo, Sarajevo
  - Uni Hospital Center Tuzla, Tuzla
- Brazil (3):
  - Santa Casa de Misericordia; de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Hospital Universitario Gaffree e Guinle, Rio de Janeiro, Rio de Janeiro
  - Hospital das Clinicas - UNICAMP, Campinas, São Paulo
- Bulgaria (4):
  - MHATNP Sv.Naum EAD; Clinic for intensive treatment of neurology diseases, Sofia
  - Fifth MHAT-Sofia AD; Neuro Dept with Vascular Unit, Sofia
  - MHAT National Cardiology Hospital, EAD; Neurology, Sofia
  - UMHAT Alexandrovska, EAD; Neurology, Sofia
- Canada (8):
  - Multiple Sclerosis Clinic, Calgary, Alberta
  - University of Alberta; Northern Alberta Trials & Research Centre, Edmonton, Alberta
  - Vancouver Hospital - UBC Hospital Site, Vancouver, British Columbia
  - The Ottawa Hospital - General Campus, Ottawa, Ontario
  - Clinique NeuroOutaouais, Gatineau, Quebec
  - Recherche Sepmus Inc., Greenfield Park, Quebec
  - Hôpital Maisonneuve - Rosemont; Recherche Clinique de Neurologie, Montreal, Quebec
  - Montreal Neurological Institute and Hospital, Montreal, Quebec
- Croatia (4):
  - General Hospital Pula, Pula
  - General Hospital Varazdin, Varaždin
  - Clinical Hospital Centre Zagreb;Clinic for Neurology, Zagreb
  - Uni Hospital Centre Dubrava, Zagreb
- Czechia (4):
  - Fakultni nemocnice Brno, Brno
  - Neurospol s.r.o., Havířov
  - Pardubicka Krajska Nemocnice; Department of Neurology, Pardubice
  - Krajska zdravotni, a. s. ? Nemocnice Teplice, o. z.; Neurologicke oddeleni, Teplice
- France (6):
  - Hopital Neurologique Pierre Wertheimer, Bron
  - Hôpital General - Service de neurologie; Service de neurologie, Dijon
  - Hôpital Saint Philibert, Lommé
  - Groupe Hospitalier Pitie-Salpetriere, Paris
  - Hôpital Maison Blanche; Service de Neurologie, Reims
  - CHU toulouse - Hôpital Purpan; Departement de Neurologie, Toulouse
- Germany (10):
  - Sankt Gertrauden Krankenhaus; Neurologisches Facharztzentrum, Berlin
  - Neurologische Praxis Bonn, Bonn
  - Universitätsklinikum Düsseldorf; Klinik für Neurologie, Düsseldorf
  - Zentrum fuer ambulante Neurologie, Essen
  - Universitaetsklinikum Frankfurt; Klinik für Neurologie, Frankfurt
  - Universitaetsklinikum Heidelberg, Heidelberg
  - Ratsapotheke Mittweida, Mittweida
  - Klinikum Grosshadern der LMU, München
  - Klinikum rechts der Isar der TU Muenchen; Neurologische Klinik und Poliklinik im Neuro-Kopf-Zentrum, München
  - Neurologische Gemeinschaftspraxis Dr. Lang, Prof. Schreiber, Dr. Krauß, Dr. Kornhuber, Ulm
- St Vincents University Hospital, Dublin, Ireland
- Italy (10):
  - Ospedale Generale Regionale F. Miulli, Acquaviva delle Fonti, Apulia
  - Ospedale Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo, Apulia
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata, Rome, Lazio
  - Policlinico Universitario Agostino Gemelli, Rome, Lazio
  - A.O. Universitaria S. Martino Di Genova, Genoa, Liguria
  - Fondazione IRCCS Istituto Neurologico Carlo Besta; Farmacia Interna, Milan, Lombardy
  - Ospedale Civile di Montichiari; Centro Sclerosi Multipla, Montichiari, Lombardy
  - Ospedale degli Infermi, Ponderano, Piedmont
  - Fond. Ist. S. Raffaele - giglio, Cefalù, Sicily
  - Azienda Ospedaliero Universitaria Ospedali Riuniti Umberto I-G.M. Lancisi-G. Salesi Di Ancona, Torrette - Ancona, The Marches
- Mexico (6):
  - Hospital Mexico Americano SC; Departamento de Electroencefalografía, Guadalajara, Jalisco
  - Mexico Centre for Clinical Research, Mexico City, Mexico CITY (federal District)
  - Clinical Research Institute, Tlalnepantla, Mexico CITY (federal District)
  - Hospital Angeles Culiacan; Neurociencias, Culiacán, Sinaloa
  - Instituto Biomedico De Investigacion A.C., Aguascalientes
  - Hospital CIMA Chihuahua; Centro de Investigación Clínicatorre de Consultoriospiso 4, Chihuahua City
- Haukeland Universitetssykehus, Bergen, Norway
- Poland (9):
  - Vitamed, Bydgoszcz
  - MA-LEK Clinical Sp. Z o.o., Katowice
  - Krakowska Akademia Neurologii Sp z o.o. Centrum Neurologii K, Krakow
  - SPZOZ Uniwersytecki Szp. Klin. nr1 im.N.Barlickiego UM;Oddzial Kliniczny Neurologii, Lodz
  - Centrum Neurologii Krzysztof Selmaj, Lodz
  - Samodz.Publi.Szpital Kliniczny; nr 4 w Lublinie, Lublin
  - Wojewodzki Specjalistyczny Szpital w Olsztynie; Oddzial Neurologiczny z Pododdzialem Udarowym, Olsztyn
  - Neuro-Care Gabriela Klodowska, Siemianowice ?l?skie
  - mMED Maciej Czarnecki, Warsaw
- Russia (8):
  - State institution of health care - Territorial Clinical Hospital, Barnaul, Altayskiy Kray
  - St. Petersburg State Medical University n.a. I.P. Pavlov; Hematology, transfusiology and transplanta, Saint Petersburg, Sankt-Peterburg
  - City Clinical Hospital#2, Pyatigorsk, Stavropol Kray
  - State autonomous institution of healthcare Inter-regional clinical and diagnostic center, Kazan', Tatarstan Republic
  - Kirov City Clinical Hospital #1; Neurology Department, Kirov
  - SBHI of Nizhny Novgorod region City Clinical Hospital #3; neurology department, Nizniy Novgorod
  - Perm SMA n.a. academ. E.A. Vagner, Perm
  - Saratov State Medical University of RosZdrav; Neurology, Saratov
- Slovakia (3):
  - MUDr. Beata Dupejova Neurologicka ambulancia s.r.o, Banská Bystrica
  - Fakultna Nemocnica Roosevelta, Banská Bystrica
  - Vseobecna nemocnica s poliklinikou Levoca a.s., Levoča
- Spain (10):
  - Institut Catala d?Oncologia Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari de Bellvitge; Servicio de Neurologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital General Univ. de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitari de Girona Dr Josep Trueta, Girona
  - Hospital General Universitario Gregorio Marañon; Servicio de Neurologia, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Clinico Universitario de Valencia; Servicio de Neurologia, Valencia
- Sweden (4):
  - Sahlgrenska Sjukhuset; Neurology, Gothenburg
  - Karolinska Universitetssjukhuset Solna Neurology, Stockholm
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
  - Norrlands Universitetssjukhus, Umeå
- Turkey (Türkiye) (8):
  - Hacettepe University Medical Faculty; Neurology, Ankara
  - Haseki Training and Research Hospital, Istanbul
  - Istanbul Universitesi - Cerrahpasa Cerrahpasa Tip Fakultesi; Noroloji Anabilim Dali, Istanbul
  - Istanbul Bilim Universty Medical Fac., Istanbul
  - Ege University Medical Faculty, Izmir
  - Kocaeli University Medical Faculty, Kocaeli
  - Ondokuz Mayis Univ. Med. Fac.; Neurology, Samsun
  - Karadeniz Tecnical Uni. Med. Fac.; Neurology, Trabzon
- Ukraine (5):
  - Mun.Med.Proph.Inst.?Chernihiv Reg.Hosp.?; Neurology Department, Chernihiv
  - City Clinical Hospital #4, Dnipropetrovsk
  - State Institution V.K. Gusak Institute of Urgent and Recover; Dep of Reconstructive Angioneurology a, Donetsk
  - Road Clinical Hospital of Donetsk Station; Neurology Department, Donetsk
  - Regional Clinical Hospital; Neurology Department, Ivano-Frankivsk
- United Kingdom (4):
  - Royal Devon and Exeter Hospital (Wonford), Exeter
  - Kings College Hospital; Neurosciences Clinical Trials Office, London
  - City General Hospital; Department of Neurology, Stoke-on-Trent
  - Morriston Hospital, Swansea

REFERENCES:
- [Derived] Kappos L, Yiu S, Reucassel J, Oh J, Granziera C, Killestein J, Bermel RA, Berge C, Kazlauskaite A, Schneble HM, Dahlke F, Cree BAC. Performance of Composite Endpoints Defining Progression Independent of Relapse Activity in Multiple Sclerosis. Ann Clin Transl Neurol. 2025 Sep;12(9):1805-1812. doi: 10.1002/acn3.70111. Epub 2025 Jul 8. PMID 40629721
- [Derived] Montobbio N, Bovis F, Signori A, Carmisciano L, Schiavetti I, Ponzano M, Tur C, Granziera C, Cagol A, Arnold DL, Kappos L, Sormani MP. Uncovering a bias in estimated treatment effects on PIRA in multiple sclerosis clinical trials. EBioMedicine. 2025 Jul;117:105802. doi: 10.1016/j.ebiom.2025.105802. Epub 2025 Jun 18. PMID 40554392
- [Derived] Kappos L, Yiu S, Dahlke F, Coetzee T, Cutter GR, Yuen S, Bonati U, Lublin FD. Composite Confirmed Disability Worsening/Progression Is a Useful Clinical Endpoint for Multiple Sclerosis Clinical Trials. Neurology. 2025 May 27;104(10):e213558. doi: 10.1212/WNL.0000000000213558. Epub 2025 Apr 21. PMID 40258203
- [Derived] Benedict RH, Kappos L, Miller A, Hartung HP, Overell J, Pei J, Dahlke F, Bernasconi C, Koendgen H, Wang Q, Bonati U, Cohan S. Cognitive effects of ocrelizumab vs interferon beta-1a in relapsing multiple sclerosis: A post hoc analysis of the OPERA I/II trials. Mult Scler Relat Disord. 2025 Mar;95:106310. doi: 10.1016/j.msard.2025.106310. Epub 2025 Feb 2. PMID 39965438
- [Derived] Muros-Le Rouzic E, Heer Y, Yiu S, Tozzi V, Braune S, van Hovell P, Bergmann A, Bernasconi C, Model F, Craveiro L; NTD study group. Five-year efficacy outcomes of ocrelizumab in relapsing multiple sclerosis: A propensity-matched comparison of the OPERA studies with other disease-modifying therapies in real-world lines of treatments. J Cent Nerv Syst Dis. 2024 Sep 13;16:11795735241260563. doi: 10.1177/11795735241260563. eCollection 2024. PMID 39290861
- [Derived] Loomis SJ, Sadhu N, Fisher E, Gafson AR, Huang Y, Yang C, Hughes EE, Marshall E, Herman A, John S, Runz H, Jia X, Bhangale T, Bronson PG. Genome-wide study of longitudinal brain imaging measures of multiple sclerosis progression across six clinical trials. Sci Rep. 2023 Aug 31;13(1):14313. doi: 10.1038/s41598-023-41099-0. PMID 37652990
- [Derived] Kolind S, Gaetano L, Assemlal HE, Bernasconi C, Bonati U, Elliott C, Hagenbuch N, Magon S, Arnold DL, Traboulsee A. Ocrelizumab-treated patients with relapsing multiple sclerosis show volume loss rates similar to healthy aging. Mult Scler. 2023 May;29(6):741-747. doi: 10.1177/13524585231162586. Epub 2023 May 6. PMID 37148240
- [Derived] Hauser SL, Bar-Or A, Weber MS, Kletzl H, Gunther A, Manfrini M, Model F, Mercier F, Petry C, Wing Q, Koendgen H, Smith T, Kappos L. Association of Higher Ocrelizumab Exposure With Reduced Disability Progression in Multiple Sclerosis. Neurol Neuroimmunol Neuroinflamm. 2023 Feb 15;10(2):e200094. doi: 10.1212/NXI.0000000000200094. Print 2023 Mar. PMID 36792367
- [Derived] Falet JR, Durso-Finley J, Nichyporuk B, Schroeter J, Bovis F, Sormani MP, Precup D, Arbel T, Arnold DL. Estimating individual treatment effect on disability progression in multiple sclerosis using deep learning. Nat Commun. 2022 Sep 26;13(1):5645. doi: 10.1038/s41467-022-33269-x. PMID 36163349
- [Derived] Arnold DL, Sprenger T, Bar-Or A, Wolinsky JS, Kappos L, Kolind S, Bonati U, Magon S, van Beek J, Koendgen H, Bortolami O, Bernasconi C, Gaetano L, Traboulsee A. Ocrelizumab reduces thalamic volume loss in patients with RMS and PPMS. Mult Scler. 2022 Oct;28(12):1927-1936. doi: 10.1177/13524585221097561. Epub 2022 Jun 7. PMID 35672926
- [Derived] Krishnan AP, Song Z, Clayton D, Gaetano L, Jia X, de Crespigny A, Bengtsson T, Carano RAD. Joint MRI T1 Unenhancing and Contrast-enhancing Multiple Sclerosis Lesion Segmentation with Deep Learning in OPERA Trials. Radiology. 2022 Mar;302(3):662-673. doi: 10.1148/radiol.211528. Epub 2021 Dec 14. PMID 34904871
- [Derived] Giovannoni G, Kappos L, de Seze J, Hauser SL, Overell J, Koendgen H, Manfrini M, Wang Q, Wolinsky JS. Risk of requiring a walking aid after 6.5 years of ocrelizumab treatment in patients with relapsing multiple sclerosis: Data from the OPERA I and OPERA II trials. Eur J Neurol. 2022 Apr;29(4):1238-1242. doi: 10.1111/ene.14823. Epub 2021 May 5. PMID 33724637
- [Derived] Hauser SL, Kappos L, Arnold DL, Bar-Or A, Brochet B, Naismith RT, Traboulsee A, Wolinsky JS, Belachew S, Koendgen H, Levesque V, Manfrini M, Model F, Hubeaux S, Mehta L, Montalban X. Five years of ocrelizumab in relapsing multiple sclerosis: OPERA studies open-label extension. Neurology. 2020 Sep 29;95(13):e1854-e1867. doi: 10.1212/WNL.0000000000010376. Epub 2020 Jul 20. PMID 32690791
- [Derived] Kappos L, Wolinsky JS, Giovannoni G, Arnold DL, Wang Q, Bernasconi C, Model F, Koendgen H, Manfrini M, Belachew S, Hauser SL. Contribution of Relapse-Independent Progression vs Relapse-Associated Worsening to Overall Confirmed Disability Accumulation in Typical Relapsing Multiple Sclerosis in a Pooled Analysis of 2 Randomized Clinical Trials. JAMA Neurol. 2020 Sep 1;77(9):1132-1140. doi: 10.1001/jamaneurol.2020.1568. PMID 32511687
- [Derived] Hauser SL, Bar-Or A, Comi G, Giovannoni G, Hartung HP, Hemmer B, Lublin F, Montalban X, Rammohan KW, Selmaj K, Traboulsee A, Wolinsky JS, Arnold DL, Klingelschmitt G, Masterman D, Fontoura P, Belachew S, Chin P, Mairon N, Garren H, Kappos L; OPERA I and OPERA II Clinical Investigators. Ocrelizumab versus Interferon Beta-1a in Relapsing Multiple Sclerosis. N Engl J Med. 2017 Jan 19;376(3):221-234. doi: 10.1056/NEJMoa1601277. Epub 2016 Dec 21. PMID 28002679

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1045 participants were screened for entry into the study. Of these, 210 participants failed screening; the main reasons were failure to meet the inclusion/exclusion criteria or unacceptable laboratory values. A total of 835 participants were enrolled in the study.
Pre-assignment Details: All participants were provided an opportunity to rollover and continue treatment and/or safety follow-up under the new extension protocol MN43964. In error, the study completion status for 5 participants was registered as 'Sponsor Termination' in the study eCRF. All 5 participants opted not to be enrolled into MN43964 and decided to pursue treatment outside the context of a clinical trial. In conclusion, the 5 participants should be considered as having completed the WA21093 study.
Groups:
- Interferon Beta-1a + Ocrelizumab Placebo: Interferon beta-1a 44 mcg SC injections three times per week (with placebo infusions matching ocrelizumab infusions every 24 weeks).
- Ocrelizumab + Interferon Beta-1a Placebo: Ocrelizumab 600 mg or matching placebo intravenous (IV) as 300 mg infusions on Days 1 and 15 for the first dose and as a single infusion of 600 mg for all subsequent infusions every 24 weeks, with placebo injections matching interferon beta-1a SC three times per week.
Period: Overall Study
Arm/Group | Interferon Beta-1a + Ocrelizumab Placebo | Ocrelizumab + Interferon Beta-1a Placebo
Started | 418 | 417
Entered OLE Period | 297 | 350
Completed | 229 | 225
Not Completed | 189 | 192
Not completed — Adverse Event | 40 | 42
Not completed — Death | 5 | 6
Not completed — Lack of Efficacy | 22 | 10
Not completed — Lost to Follow-up | 15 | 12
Not completed — Non-Compliance | 3 | 7
Not completed — Non-Compliance With Study Drug | 1 | 1
Not completed — Other | 30 | 33
Not completed — Physician Decision | 11 | 16
Not completed — Pregnancy | 6 | 4
Not completed — Protocol Violation | 1 | 2
Not completed — Study Terminated By Sponsor | 3 | 2
Not completed — Withdrawal by Subject | 51 | 54
Not completed — Missing | 1 | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all randomized participants in the study.
Groups:
- Interferon Beta-1a + Ocrelizumab Placebo (Double Blind Period): Interferon beta-1a 44 mcg SC injections three times per week (with placebo infusions matching ocrelizumab infusions every 24 weeks).
- Ocrelizumab + Interferon Beta-1a Placebo (Double Blind Period): Ocrelizumab 600 mg or matching placebo intravenous (IV) as 300 mg infusions on Days 1 and 15 for the first dose and as a single infusion of 600 mg for all subsequent infusions every 24 weeks, with placebo injections matching interferon beta-1a SC three times per week.
- Total: Total of all reporting groups
Arm/Group | Interferon Beta-1a + Ocrelizumab Placebo (Double Blind Period) | Ocrelizumab + Interferon Beta-1a Placebo (Double Blind Period) | Total
Number analyzed (Participants) | 418 | 417 | 835
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.4 (9.0) | 37.2 (9.1) | 37.3 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 280 | 271 | 551
  Male | 138 | 146 | 284

OUTCOME MEASURES:

1. Primary Outcome: Annualized Relapse Rate (ARR) in Participants With Relapsing Multiple Sclerosis (MS) at 96 Weeks In Double Blind Period
Description: ARR was protocol-defined and calculated as the total number of relapses for all participants in the treatment group divided by the total participant-years of exposure to that treatment.
Time Frame: Week 96
Population: Intent-to-treat (ITT) population included all randomized participants in the study.
Measure: Number (95% Confidence Interval); unit: relapses/participant year of treatment
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 418 | 417
relapses/participant year of treatment | 0.290 [0.234 to 0.361] | 0.155 [0.121 to 0.198]
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Adjusted by Geographical Region (US vs. Rest of World) and baseline EDSS (<4.0 vs. >=4.0); Test type: Superiority or Other; p < 0.0001, Negative Binomial Model; Rate Ratio = 0.532, 95% CI 2-sided [0.397 to 0.714] — Rate ratio was calculated as Ocrelizumab ARR/Interferon beta-1a 44 mcg SC ARR

2. Secondary Outcome: Time to Onset of Confirmed Disability Progression (CDP) for at Least 12 Weeks During the Double-Blind Treatment Period
Description: Disability progression was defined as an increase in the Expanded Disability Status Scale (EDSS) score of: A) >=1.0 point from the baseline EDSS score when the baseline score was less than or equal to (<=) 5.5 B) >=0.5 point from the baseline EDSS score when the baseline score was >5.5 The EDSS scale ranges from 0 (normal neurological exam) to 10 (death due to multiple sclerosis). This outcome measure was considered confirmatory only when results of both studies WA21092 and WA21093 were combined. Disability progression was considered confirmed when the increase in the EDSS was confirmed at a regularly scheduled visit at least 12 weeks after the initial documentation of neurological worsening. Participants who had initial disability progression with no confirmatory EDSS assessment and who were on treatment at time of clinical cut-off date were censored at the date of their last EDSS assessment.
Time Frame: Week 104
Population: ITT population included all randomized participants in the study.
Measure: Median (Full Range); unit: weeks
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 418 | 417
weeks | NA [0 to 102] — Median of time to onset of CDP was not achieved due to low number of participants with events. The full-range values are censored observations. | NA [0 to 104] — Median of time to onset of CDP was not achieved due to low number of participants with events. The lower-limit value is a censored observation.
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Time to onset of CDP at week 12; Test type: Superiority or Other; p = 0.0169, Log Rank; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.42 to 0.92]

3. Secondary Outcome: Number of T1 Gadolinium (Gd)-Enhancing Lesions as Detected by Brain Magnetic Resonance Imaging (MRI) During the Double-Blind Treatment
Description: The total number of T1 gadolinium-enhancing lesions for all participants in the treatment group was calculated as the sum of the individual number of lesions at Weeks 24, 48, and 96.
Time Frame: Baseline up to week 96
Population: ITT population included all randomized participants in the study.
Measure: Number; unit: lesions
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 418 | 417
lesions | 465 | 21
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Test type: Superiority or Other; p < 0.0001, Negative Binomial Model; Adjusted rate ratio = 0.051, 95% CI [0.029 to 0.089] — Adjusted by baseline T1 Gd lesion (present or not), baseline EDSS (<4.0 vs. >=4.0) and geographical region (US vs. rest-of-world). Adjusted rate ratio was calculated as Ocrelizumab adjusted rate/Interferon beta-1a 44 mcg SC adjusted rate

4. Secondary Outcome: Number of New, and/or Enlarging T2 Hyperintense Lesions as Detected by Brain Magnetic Resonance Imaging (MRI) During the Double Blind Treatment
Description: The total number of new and/or enlarging T2 lesions for all participants in the treatment group was calculated as the sum of the individual number of lesions at Weeks 24, 48, and 96.
Time Frame: Baseline up to week 96
Population: ITT population included all randomized participants in the study.
Measure: Number; unit: lesions
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 418 | 417
lesions | 2103 | 380
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Test type: Superiority or Other; p < 0.0001, Negative Binomial Model; Adjusted rate ratio = 0.171, 95% CI [0.130 to 0.225] — Adjusted by baseline T2 lesion count, baseline EDSS (<4.0 vs. >=4.0) and geographical region (US vs. rest-of-world). Adjusted rate ratio was calculated as Ocrelizumab adjusted rate/Interferon beta-1a 44 mcg SC adjusted rate

5. Secondary Outcome: Percentage of Participants With Confirmed Disability Improvement (CDI) for at Least 12 Weeks In Double Blind Period
Description: Disability improvement was assessed only for the subgroup of participants with a baseline EDSS score of >= 2.0. It was defined as a reduction in EDSS score of: A) >=1.0 from the baseline EDSS score when the baseline score was >=2 and <=5.5 B) >= 0.5 when the baseline EDSS score > 5.5. The EDSS scale ranges from 0 (normal neurological exam) to 10 (death due to multiple sclerosis). This outcome measure was considered confirmatory only when results of both studies WA21092 and WA21093 were combined.
Time Frame: Week 96
Population: ITT population included all randomized participants in the study. Here, number of participants analyzed signifies number of participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 308 | 318
percentage of participants | 18.83 [14.62 to 23.65] | 21.38 [17.01 to 26.30]
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Test type: Superiority or Other; p = 0.4019, CMH Chi-Squared test (stratified); Stratified by Geographical Region (US vs. Rest of World) and baseline EDSS (<4.0 vs. >=4.0); Relative risk (stratified) = 1.14, 95% CI 2-sided [0.84 to 1.56]

6. Secondary Outcome: Time to Onset of Confirmed Disability Progression (CDP) for at Least 24 Weeks During the Double-Blind Treatment Period
Description: Disability progression was defined as an increase in the Expanded Disability Status Scale (EDSS) score of: A) >=1.0 point from the baseline EDSS score when the baseline score was less than or equal to (<=) 5.5 B) >=0.5 point from the baseline EDSS score when the baseline score was >5.5 The EDSS scale ranges from 0 (normal neurological exam) to 10 (death due to multiple sclerosis). This outcome measure was considered confirmatory only when results of both studies WA21092 and WA21093 were combined. Disability progression was considered confirmed when the increase in the EDSS was confirmed at a regularly scheduled visit at least 24 weeks after the initial documentation of neurological worsening. Participants who had initial disability progression with no confirmatory EDSS assessment and who were on treatment at time of clinical cut-off date were censored at the date of their last EDSS assessment.
Time Frame: Week 104
Population: ITT population included all randomized participants in the study.
Measure: Median (Full Range); unit: weeks
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 418 | 417
weeks | NA [0 to 102] — Median of time to onset of CDP was not achieved due to low number of participants with events. The full-range values are censored observations. | NA [0 to 104] — Median of time to onset of CDP was not achieved due to low number of participants with events. The full-range values are censored observations.
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Time to onset of CDP at week 24; Test type: Superiority or Other; p = 0.037, Log Rank; Hazard Ratio (HR) = 0.63, 95% CI 2-sided [0.40 to 0.98]

7. Secondary Outcome: Number of T1 Hypointense Lesions During the Double-Blind Treatment
Description: The total number of new T1-Hypo-Intense Lesions (Chronic Black Holes) for all participants in the treatment group was calculated as the sum of the individual number of new lesions at Weeks 24, 48, and 96.
Time Frame: Baseline up to week 96
Population: ITT population included all randomized participants in the study.
Measure: Number; unit: lesions
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 418 | 417
lesions | 1484 | 567
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Test type: Superiority or Other; p < 0.0001, Negative Binomial Model; Adjusted rate ratio = 0.357, 95% CI [0.272 to 0.47] — Adjusted by baseline T1-hypointense lesion count, baseline EDSS (<4.0 vs. >=4.0) and geographical region (US vs. rest-of-world). Adjusted rate ratio was calculated as Ocrelizumab adjusted rate/Interferon beta-1a 44 mcg SC adjusted rate

8. Secondary Outcome: Change From Baseline in Multiple Sclerosis Functional Composite (MSFC) Score to Week 96 In Double Blind Period
Description: MSFC score consists of: A) Timed 25-Foot walk; B) 9-Hole Peg Test (9-HPT); and C) Paced Auditory Serial Addition Test (PASAT-3 version). The MSFCS is based on the concept that scores for these three dimensions (arm, leg, and cognitive function) are combined to create a single score (the MSFC) that can be used to detect change over time in a group of participants with MS. Since the three primary measures differ in what they actually measure, a common composite score for the three different measures i.e., Z- score was selected for the purpose. MSFC Score = {Z arm, average + Z leg, average + Z cognitive} / 3.0. The results from each of these three tests are transformed into Z-scores and averaged to yield a composite score for each participant at each time point. A score of +1 indicates that, on average, an individual scored 1 standard deviation (SD) better than the reference population and a score of -1 indicates that an individual scored 1 SD worse than the reference population.
Time Frame: Baseline, Week 96
Population: ITT population included all randomized participants in the study. Here, n signifies the number of participants evaluable at specified time points.
Measure: Mean (Standard Error); unit: Z-score
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 418 | 417
Z-score
  Unadjusted Baseline mean (n= 342, 358) | -0.001 (0.033) | 0.026 (0.034)
  Adjusted Week 96 mean (n= 269, 308) | 0.169 (0.029) | 0.276 (0.028)
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Test type: Superiority or Other; p = 0.004, mixed-effect model of repeated measures; Estimates are from analysis based on mixed-effect model of repeated measures (MMRM) using unstructured covariance matrix; Difference in Adjusted Means = 0.107, 95% CI 2-sided [0.034 to 0.180], Standard Error of Mean 0.037 — Difference in adjusted means was calculated as Ocrelizumab adjusted mean at Week 96/ Interferon beta-1a 44 mcg SC adjusted mean at Week 96

9. Secondary Outcome: Percent Change in Brain Volume as Detected by Brain Magnetic Resonance Imaging (MRI) From Week 24 to Week 96 In Double Blind Period
Description: Brain volume was recorded as an absolute "normalized" value at the baseline visit then recorded at subsequent visits as a percentage change relative to the absolute value at the baseline visit. Therefore, brain volume at Week 24 was calculated as the brain volume at the baseline visit multiplied by 1 + ([percentage change in brain volume from baseline visit to Week 24]/100). Estimates are from analysis based on mixed-effect model of repeated measures (MMRM) using unstructured covariance matrix: Percentage Change = Brain Volume at Week 24 + Geographical Region (US vs. ROW) + Baseline EDSS (< 4.0 vs. >= 4.0) + Week + Treatment + Treatment*Week (repeated values over Week) + Brain Volume at Week 24*Week. The EDSS scale ranges from 0 (normal neurological exam) to 10 (death due to multiple sclerosis).
Time Frame: From week 24 up to week 96
Population: as for outcome 5
Measure: Mean (Standard Error); unit: percent change
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 259 | 287
percent change | -0.75 (0.051) | -0.638 (0.049)
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Test type: Superiority or Other; p = 0.09, mixed-effect model of repeated measures; [statistical method as in outcome 8, analysis 1]; Difference in Adjusted Means = 0.112, 95% CI 2-sided [-0.018 to 0.241], Standard Error of Mean 0.066 — Difference in the rate of brain volume loss: 14.9%. Difference in adjusted means was calculated as Ocrelizumab adjusted mean at Week 96/ Interferon beta-1a 44 mcg SC adjusted mean at Week 96

10. Secondary Outcome: Change From Baseline in Short Form Health Survey-36 (SF-36) Physical Component Summary (PCS) Score at Week 96 In Double Blind Period
Description: The SF-36 is a multi-purpose, short-form health survey with 36 questions. It yields an 8-scale profile of functional health and well-being scores (domains) as well as psychometrically based physical and mental health summary measures. The SF-36 taps 8 health concepts: physical functioning, bodily pain, physical role functioning, emotional role functioning, emotional well-being, social functioning, vitality, and general health perceptions. The 8 scales are further summarized to 2 distinct higher-ordered clusters: the PCS and mental composite t-score (MCS). The range for all 8 domains as well as for the composite t- scores is from 0 to 100 with 100 as best possible health status and 0 as worst health status.
Time Frame: Baseline, Week 96
Population: Descriptive statistics at baseline include participants with assessment at baseline and at least one post- baseline value. ITT population included all randomized participants in the study. Here, n signifies the number of participants evaluable at specified time points.
Measure: Mean (Standard Error); unit: t-score
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 418 | 417
t-score
  Unadjusted Baseline mean (n= 319, 355) | 44.552 (0.544) | 44.307 (0.541)
  Adjusted mean change at week 96(n=276, 315) | -0.833 (0.472) | 0.326 (0.444)
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Test type: Superiority or Other; p = 0.0404, mixed-effect model of repeated measures; Estimates are from analysis based on mixed-effect model of repeated measures using unstructured covariance matrix; Difference in Adjusted Means = 1.159, 95% CI 2-sided [0.051 to 2.268], Standard Error of Mean 0.564 — [estimate comment as in outcome 8, analysis 1]

11. Secondary Outcome: Percentage of Participants Who Have No Evidence of Disease Activity (NEDA) up to Week 96 In Double Blind Period
Description: NEDA was defined only for participants with a baseline EDSS score >=2.0. The EDSS scale ranges from 0 (normal neurological exam) to 10 (death due to multiple sclerosis). Participants who completed the 96- week treatment period were considered as having evidence of disease activity if at least one protocol- defined relapse (PDR), a confirmed disability progression (CDP) event or at least one MRI scan showing MRI activity (defined as Gd-enhancing T1 lesions, or new or enlarging T2 lesions) was reported during the 96-week treatment period, otherwise the participant was considered as having NEDA.
Time Frame: Week 96
Population: ITT population included all randomized participants in the study. Here, number of participants analysed signifies number of participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 270 | 289
percentage of participants | 24.1 [19.1 to 29.6] | 43.9 [38.1 to 49.9]
Statistical Analysis 1: Comparison: Interferon Beta-1a 44 mcg SC vs Ocrelizumab; Test type: Superiority or Other; p < 0.0001, CMH Chi-Squared test (stratified); Analyzed using CMH test, stratified by Geographical Region (US vs. rest-of-world) and baseline EDSS (<4.0 vs. >=4.0); Relative risk (stratified) = 1.81, 95% CI 2-sided [1.41 to 2.32]

12. Secondary Outcome: Number of Participants With Adverse Events (AEs)
Description: AEs included infusion related reactions (IRRs) and serious MS relapses, but excluded non-serious MS relapses. Serious Adverse Events (SAEs) included serious MS relapses and serious IRRs.
Time Frame: Baseline up to Week 96
Population: The safety population included all participants who received any study drug.
Measure: Number; unit: participants
Groups:
- Interferon Beta-1a + Placebo (Open Label Extension); Ocrelizumab + Placebo (Open Label Extension): During the OLE phase, all participants received ocrelizumab 600-mg IV infusion every 24 weeks.
Arm/Group | Interferon Beta-1a + Ocrelizumab Placebo (Double Blind Period) | Ocrelizumab + Interferon Beta-1a Placebo (Double Blind Period) | Interferon Beta-1a + Placebo (Open Label Extension) | Ocrelizumab + Placebo (Open Label Extension)
Number analyzed (Participants) | 417 | 417 | 297 | 350
participants
  Adverse Events | 357 | 360 | 281 | 333
  Serious Adverse Events | 40 | 29 | 71 | 121

13. Secondary Outcome: Exposure to Ocrelizumab (Area Under the Concentration - Time Curve, AUC) In Double Blind Period
Description: AUC represents total drug exposure for one dosing interval after the 4th dose.
Time Frame: Pre-infusion at Weeks 1, 24, 48, 72; and 30 minutes post-infusion at Week 72; at any time during Weeks 84 and 96
Population: The pharmacokinetics (PK) population included all participants in the ocrelizumab group who had at least 1 measurable concentration value.
Measure: Mean (Standard Deviation); unit: micrograms per milliter*day
Arm/Group | Ocrelizumab
Number analyzed (Participants) | 389
micrograms per milliter*day | 3513 (955)

14. Secondary Outcome: Number of Participants With Anti-Drug Antibodies (ADAs) to Ocrelizumab In Double Blind Period
Description: Number of participants positive for anti-drug antibodies (ADAs) to ocrelizumab is the number of post- baseline evaluable participants determined to have treatment-induced ADA or treatment-enhanced ADA during the study period.
Time Frame: Baseline up to Week 96
Population: Baseline evaluable participants with an ADA assay result from a baseline sample(s). The safety population included all participants who received any study drug. Here, n signifies the number of participants evaluable at the specified time points.
Measure: Number; unit: participants
Arm/Group | Interferon Beta-1a 44 mcg SC | Ocrelizumab
Number analyzed (Participants) | 417 | 417
participants
  Positive sample at baseline (n= 407, 402) | 2 | 4
  Positive for ADA post-baseline (n= 403, 405) | 5 | 2

ADVERSE EVENTS:
Time Frame: Baseline to approximately 588 weeks
Description: The safety population included all participants who received any study drug.
Groups:
- Interferon Beta-1a + Ocrelizumab Placebo (Double Blind): Interferon beta-1a 44 mcg SC injections three times per week (with placebo infusions matching ocrelizumab infusions every 24 weeks).
- Ocrelizumab + Interferon Beta-1a Placebo (Double Blind): Ocrelizumab 600 mg or matching placebo intravenous (IV) as 300 mg infusions on Days 1 and 15 for the first dose and as a single infusion of 600 mg for all subsequent infusions every 24 weeks, with placebo injections matching interferon beta-1a SC three times per week.
- Interferon Beta-1a + Ocrelizumab Placebo (Double Blind) Ocrelizumab (Open Label): In DB phase participants received Interferon Beta-1a and Ocrelizumab Placebo. During the OLE phase, all participants received ocrelizumab 600-mg IV infusion every 24 weeks.
- Ocrelizumab + Interferon Beta-1a Placebo (Double Blind) Ocrelizumab (Open Label): In DB phase participants received Ocrelizumab + Interferon Beta-1a Placebo. During the OLE phase, all participants received ocrelizumab 600-mg IV infusion every 24 weeks.
Arm/Group | Interferon Beta-1a + Ocrelizumab Placebo (Double Blind) | Ocrelizumab + Interferon Beta-1a Placebo (Double Blind) | Interferon Beta-1a + Ocrelizumab Placebo (Double Blind) Ocrelizumab (Open Label) | Ocrelizumab + Interferon Beta-1a Placebo (Double Blind) Ocrelizumab (Open Label)
All-Cause Mortality (participants affected / at risk) | 1/417 | 1/417 | 5/297 | 6/350
Serious Adverse Events (participants affected / at risk) | 40/417 | 29/417 | 71/297 | 121/350
Other Adverse Events (participants affected / at risk) | 357/417 | 360/417 | 266/297 | 317/350
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon Beta-1a + Ocrelizumab Placebo (Double Blind) (N=417) | Ocrelizumab + Interferon Beta-1a Placebo (Double Blind) (N=417) | Interferon Beta-1a + Ocrelizumab Placebo (Double Blind) Ocrelizumab (Open Label) (N=297) | Ocrelizumab + Interferon Beta-1a Placebo (Double Blind) Ocrelizumab (Open Label) (N=350)
ANAEMIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SPLENIC VEIN THROMBOSIS (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SPONTANEOUS HAEMATOMA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TRISOMY 21 (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GOITRE (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
THYROIDITIS SUBACUTE (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CATARACT (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RETINAL DETACHMENT (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
APPENDICITIS NONINFECTIVE (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CROHN'S DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DIVERTICULUM (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENTEROVESICAL FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROINTESTINAL INFLAMMATION (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ILEUS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ILEUS PARALYTIC (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
MECHANICAL ILEUS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OESOPHAGITIS (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PANCREATITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PANCREATITIS ACUTE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SMALL INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DEATH (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BILE DUCT STENOSIS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (3)
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2)
CHOLELITHIASIS (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
HEPATITIS ACUTE (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEPATITIS FULMINANT (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LIVER DISORDER (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HAEMOPHAGOCYTIC LYMPHOHISTIOCYTOSIS (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACUTE HEPATITIS C (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ACUTE SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
ANAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
APPENDICITIS (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
ATYPICAL PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CELLULITIS PHARYNGEAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CHOLECYSTITIS INFECTIVE (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CHRONIC SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 9 (9) | 13 (13)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 13 (13) | 23 (24)
CYSTITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
ENCEPHALITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ENTEROCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENTEROVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FURUNCLE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTRITIS VIRAL (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
INJECTION SITE CELLULITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LYME DISEASE (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MASTOIDITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MENINGITIS ASEPTIC (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MENINGITIS VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ORCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTITIS MEDIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PARASITIC GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PASTEURELLA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PELVIC INFLAMMATORY DISEASE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
PERIRECTAL ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PHARYNGITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 2 (2) | 1 (1) | 6 (7) | 15 (15)
PNEUMONIA ASPIRATION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
PNEUMONIA BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PNEUMONIA HAEMOPHILUS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA VIRAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
POSTOPERATIVE WOUND INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (4) | 0 (0)
PYELONEPHRITIS (Infections and infestations) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
PYELONEPHRITIS ACUTE (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PYURIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKIN INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
STAPHYLOCOCCAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 4 (5) | 3 (3)
UROSEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VASCULAR DEVICE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
VIRAL INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
VIRAL PERICARDITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VIRAL SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ACETABULUM FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ALCOHOL POISONING (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
ANASTOMOTIC LEAK (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRAIN CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CARTILAGE INJURY (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CLAVICLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EPICONDYLITIS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FIBULA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FRACTURE DISPLACEMENT (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAND FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INCISIONAL HERNIA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (2) | 0 (0)
JAW FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
JOINT INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LOWER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MENISCUS INJURY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
MULTIPLE INJURIES (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SKULL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SPINAL CORD INJURY CAUDA EQUINA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SUBDURAL HAEMATOMA (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
TOXICITY TO VARIOUS AGENTS (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TRAUMATIC INTRACRANIAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HYPOPROTEINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
IMPAIRED INSULIN SECRETION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTERVERTEBRAL DISC DISORDER (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (4) | 1 (1)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
SYNOVIAL CYST (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
VERTEBRAL OSTEOPHYTE (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLADDER CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
CHONDROSARCOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
FIBROADENOMA OF BREAST (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTRADUCTAL PROLIFERATIVE BREAST LESION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
METASTATIC MALIGNANT MELANOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OVARIAN GERM CELL TERATOMA BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TESTIS CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
THYROID ADENOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TUMOUR RUPTURE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CEREBRAL INFARCTION (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COGNITIVE DISORDER (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EPILEPSY (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
FACIAL PARALYSIS (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
HEAD DISCOMFORT (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYDROCEPHALUS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LUMBOSACRAL RADICULOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MULTIPLE SCLEROSIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
MULTIPLE SCLEROSIS PSEUDO RELAPSE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 2 (2) | 1 (1) | 2 (2) | 2 (2)
NEUROLOGICAL SYMPTOM (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
OPTIC NEURITIS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRESYNCOPE (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RADICULOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
SEIZURE (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
SPINAL CORD COMPRESSION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TRIGEMINAL NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABORTION SPONTANEOUS (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
BREECH PRESENTATION (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
APATHY (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COMPLETED SUICIDE (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
CONVERSION DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
DEPRESSION SUICIDAL (Psychiatric disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
DEPRESSIVE DELUSION (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MAJOR DEPRESSION (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MENTAL STATUS CHANGES (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
PSYCHOTIC DISORDER (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
STRESS (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SUICIDAL IDEATION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
SUICIDE ATTEMPT (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
CALCULUS BLADDER (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEPHRITIS (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
URETHRAL CYST (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ADENOMYOSIS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COITAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSMENORRHOEA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ENDOMETRIOSIS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HEAVY MENSTRUAL BLEEDING (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
MENOMETRORRHAGIA (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OVARIAN CYST (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
UTERINE POLYP (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
ACUTE RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HYPERSENSITIVITY PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LARYNGEAL OEDEMA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PARANASAL SINUS INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
PULMONARY INFARCTION (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TONSILLAR INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TRACHEAL STENOSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
STERILISATION (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEEP VEIN THROMBOSIS (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERIPHERAL VENOUS DISEASE (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VARICOSE VEIN (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Interferon Beta-1a + Ocrelizumab Placebo (Double Blind) (N=417) | Ocrelizumab + Interferon Beta-1a Placebo (Double Blind) (N=417) | Interferon Beta-1a + Ocrelizumab Placebo (Double Blind) Ocrelizumab (Open Label) (N=297) | Ocrelizumab + Interferon Beta-1a Placebo (Double Blind) Ocrelizumab (Open Label) (N=350)
FATIGUE (General disorders) | 39 (52) | 44 (57) | 39 (55) | 50 (70)
INFLUENZA LIKE ILLNESS (General disorders) | 92 (106) | 23 (25) | 15 (17) | 26 (28)
PYREXIA (General disorders) | 25 (34) | 15 (18) | 20 (22) | 34 (53)
BRONCHITIS (Infections and infestations) | 13 (15) | 22 (28) | 25 (33) | 57 (85)
INFLUENZA (Infections and infestations) | 20 (25) | 24 (30) | 38 (54) | 55 (66)
NASOPHARYNGITIS (Infections and infestations) | 41 (60) | 80 (128) | 65 (120) | 96 (327)
SINUSITIS (Infections and infestations) | 20 (25) | 27 (35) | 34 (46) | 47 (84)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 53 (89) | 65 (109) | 86 (267) | 107 (325)
URINARY TRACT INFECTION (Infections and infestations) | 39 (48) | 43 (74) | 79 (212) | 96 (257)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 50 (64) | 158 (271) | 97 (177) | 63 (168)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 27 (33) | 22 (28) | 44 (57) | 53 (68)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 18 (19) | 28 (31) | 44 (65) | 48 (61)
MYALGIA (Musculoskeletal and connective tissue disorders) | 27 (30) | 12 (13) | 17 (29) | 15 (16)
HEADACHE (Nervous system disorders) | 71 (106) | 60 (88) | 49 (73) | 68 (95)
DEPRESSION (Psychiatric disorders) | 31 (34) | 29 (32) | 35 (40) | 38 (45)
INSOMNIA (Psychiatric disorders) | 23 (24) | 23 (28) | 22 (25) | 21 (26)
CONSTIPATION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 13 (15) | 20 (22)
DIARRHOEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 19 (32) | 30 (37)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 17 (25) | 22 (25)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 66 (79) | 96 (120)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 15 (26) | 21 (37)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 15 (17) | 24 (28)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 7 (7) | 21 (28)
ORAL HERPES (Infections and infestations) | 0 (0) | 0 (0) | 10 (16) | 21 (50)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 11 (11) | 23 (28)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 16 (20) | 25 (41)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 6 (7) | 18 (19)
CONTUSION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 15 (15) | 15 (21)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 18 (19) | 23 (27)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 14 (20) | 20 (25)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 15 (28) | 19 (27)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 15 (16) | 16 (20)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 33 (60) | 42 (60)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 21 (41) | 24 (38)
MULTIPLE SCLEROSIS RELAPSE (Nervous system disorders) | 0 (0) | 0 (0) | 70 (150) | 82 (157)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 21 (27) | 26 (39)
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 26 (43) | 58 (89)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 17 (22) | 21 (25)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 23 (28) | 25 (30)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 14 (15) | 26 (27)
INJECTION SITE ERYTHEMA (General disorders) | 55 (59) | 1 (1) | 0 (0) | 0 (0)
INJECTION SITE REACTION (General disorders) | 28 (28) | 2 (2) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 23 (27) | 17 (19) | 0 (0) | 0 (0)
MIGRAINE (Nervous system disorders) | 0 (0) | 0 (0) | 9 (19) | 20 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/33/NCT01412333/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-20): https://cdn.clinicaltrials.gov/large-docs/33/NCT01412333/SAP_001.pdf